


Research legislation: Ordinance on human research with the exception of Clinical trials (HRO).

Type of Research Project: Research project involving human subjects

Risk Categorisation: Category A in accordance with the ordinance HRO Art.7

SAV-IOL SA, Falaises 74, 2000 Neuchâtel, Switzerland CHE-114.948.271

Investigator

Institution Jules Gonin Eye Hospital / Fondation Asile des Aveugles Avenue de France 15, Lausanne, Switzerland CHE-109.382.412

| Name | Function | | Signature |
|---|---|---|---|
| Dr. Max Boysset | CEO SAV-IOL SA -<br>Sponsor | ot nov laro | # |
| Sabrina Sinkovic | Quality Manager -<br>Sponsor | 05-NOV-2020 | Sinlerie |
| Alexandre Pascarella | COO - Sponsor | 04-Nov-702 | Fully |
| Dr Kate Hashemi | Principal Investigator | 13 NOV 2020 | Krahein |




### **Table of protocol changes**

| Versions | Dates | Changes |
|---|---|---|
| V1 | 20 DEC 2018 | Initial version |
| V2 | 23 JAN 2019 | Address and responsibilities - Precisions in number |
| | | of patients, follow up and monitoring – Budget |
| V3 | 20 MAY 2019 | Budget update - Study duration update - Precisions |
| | | in chapters 1.2, 1.3, 2.2, 4.3, 5, 7.1 & 7.2 |
| V4 | 15 JUL 2019 | Precisions about data collection and analysis 7.1, 7.2 |
| V5 | 15 OCT 2019 | Precisions in data collection in chap. 4.3 and addition |
| | | of visits summary table in chap 4.4, review of |
| | | adverse events definitions and procedure in chap 6. |
| V6 | 06-DEC-2019 | Corrections following investigators review in cha |
| | | 1.3, 2.2, 2.6, 3.2, 4.3.2, 4.3.3, 4.4, 4.7, 6.1, 7.1, 7.3 |
| | | and 8.1. Update of chap. 11. |
| V7 | 28-JAN-2020 | Update of signatories |
| V8 | 24-FEB-2020 | Extension of inclusion period |
| | | New principal investigator (2.3, 6.2.1, 12) |
| | | Corrections following Ethic committee review: |
| | | Update of first page with research legislation type as |
| V9 | 04-NOV-2020 | HRO and risk category A, 3.1, 3.2, 4.3, 4.4 (update |
| VS | 04-1107-2020 | of table of collected data), 7.1, 7.2, 7.3, 8.3, 8.4, 8.5, |
| | | 8.7, 9, 11 |
| | | In chap 8.3: Replacement of EU medical devices |
| | | directive 93/42/EEC by the Regulation 2017/745. |




### **TABLE OF CONTENTS**

#### Contents 1.1 Background......5 1.2 1.3 Benefit risk ratio 6 2.1 2.2 Study design .......8 2.3 2.4 2.5 Facilities 8 2.6 SELECTION OF PATIENTS ......9 3.1 Patient selection method 9 3.2 Selection Criteria 9 3.3 Non-inclusion criteria 10 4.1 4.2 Treatment 11 4.3 4.3.1 4.3.2 4.3.3 4.3.4 Data collected after surgery at day 1:......11 4.3.5 Evaluation schedule 12 4.5 4.6 4.7 ASSESSMENT METHODS.......15 6 6.1




| SS ADVANCED VISION |
|--------------------|
| INTRAOCULAR LENS |

| | 6.1 | .1 Definition and classification of adverse events: | 16 |
|----|-------|-------------------------------------------------------|----|
| | 6.1 | .2 Causal relationship of adverse event | 17 |
| | 6.1 | .3 Severity of the adverse event | 17 |
| | 6.2 | Procedures | 17 |
| | 6.2 | .1 Serious adverse events and pregnancy | 17 |
| | 6.2 | .2 Other adverse events | 18 |
| 7 | DA | TA COLLECTION AND ANALYSIS | 18 |
| | 7.1 | Data collection | 18 |
| | 7.2 | Statistical analysis | 18 |
| | 7.3 | Required sample size | 19 |
| 8 | ET | HICAL AND LEGAL CONSIDERATIONS | 20 |
| | 8.1 | Medical-regulatory framework of the study | 20 |
| | 8.2 | Investigator's responsibilities | 20 |
| | 8.3 | Ethics committee | 20 |
| | 8.4 | Patient information leaflet and informed consent form | 21 |
| | 8.5 | Protection of personal data | 22 |
| | 8.6 | Premature discontinuation of the study | 22 |
| | 8.7 | Record keeping / archiving. | 22 |
| | 8.8 | Quality assurance - audit procedures | 23 |
| 9 | US | E OF RESULTS | 23 |
| 10 | ) FIN | NANCIAL ASPECTS | 23 |
| | 10.1 | Investigator fees | 23 |
| | 10.2 | Sponsor fees | 23 |
| | 10.3 | Additional costs | 24 |
| 11 | I SC | HEDULE | 25 |
| 12 | 2 SIC | GNATURES | 25 |




#### 1 INTRODUCTION

### 1.1 Background

Refractory function in patients with a cataract is mainly restored by implanting intraocular lenses (IOL) destined to replace the crystalline lens. While new surgical techniques for removing the crystalline lens have been developed, these lenses have been considerably perfected to resemble the natural crystalline lens as closely as possible.

Since December 2015, SAV-IOL SA got the CE marking with lenses which have the potential to obtain the best results in terms of visual acuity and comfort. Both are benefiting from the Instant Focus © technology (legal manufacturer SAV-IOL-SA www.sav-iol.com)

- The lens InFo is a refractive/diffractive hybrid lens characterized by extended depth of focus to guarantee satisfactory vision, regardless of focal length and light conditions. This benefit is particularly apparent for intermediate vision, significantly improved relative to multifocal optics that only allow focus on objects in near and far vision, without any usual adverse events met with that multi/polyfocal lenses
- The lens Lucidis is a refractive lens with an extended depth of focus to get satisfactory vision, regardless of focal length and light conditions. This benefit is particularly apparent for far vision, with additional view for near and intermediate vision. Lucidis is proposed in 2 sizes: 10.8 mm (Lucidis 108M) & 12.4 mm (Lucidis 124M) diameter, containing the same optical size (6.0 mm diameter).

## 1.2 Study Rationale

The objectives of the study is to evaluate efficacy and long-term safety of the Lucidis lens. Through this PMCF (post marketing clinical follow-up), the objective is to obtain an up-to-date clinical evaluation of the medical device thus supplementing data from experimental trials. Clinical and functional changes in the implanted eyes among a patient population in which the opaque crystalline lens resulting from cataract was removed and replaced by a Lucidis IOL will be described.

The objectives involve both evaluation of changes in ocular function in terms of visual acuity and comfort and listing possible complications of surgery and adverse reactions.




Study primary objectives – measure of:

- Far Best Corrected Visual Acuity in photopic conditions
- Near, intermediate and far Uncorrected visual acuity in photopic conditions
- Far Best Corrected Visual Acuity in mesopic conditions
- Near, intermediate and far Uncorrected visual acuity in mesopic conditions

Study secondary objectives - measure of:

- Contrast sensitivity in photopic conditions
- Contrast sensitivity in mesopic conditions
- Adverse reactions.

#### 1.3 Benefit risk ratio

Contraindications for intraocular lens are previous pathologies or physiological conditions, which may be aggravated by the lens, or in cases where the lens may interfere with the possibility of examining or treating diseases.

- Acute eye diseases or external or internal infection
- · Fuchs' proliferative diabetic retinopathy
- Severe corneal dystrophy
- High myopia
- Chronic or recurrent severe uveitis
- Severe optic nerve atrophy
- Congenital bilateral cataracts or non-age-related cataract
- Glaucoma
- Choroidal hemorrhage
- Color vision deficiencies
- Irregular corneal astigmatism
- Extremely shallow anterior chamber
- Severe Microphthalmos or Macrophthalmos
- Aniridia
- Retinal Detachment
- Macular degeneration
- Micropupil

Severe complications during surgery might be:

- Choroidal hemorrhage
- Vitreous loss




Adverse reactions and complications due to, or following surgery and, implantation of any intraocular lens may include, but are not limited to:

- Increased Astigmatism
- Corneal Decompensation
- Vitritis
- Loss of Best Spectacle Corrected Visual Acuity
- Lens Dislocation
- Lens Vault
- Anterior Subcapsular Cataract
- Macular Edema
- Iritis
- Decentration/Rotation of the InFo lens
- Non-reactive Pupil
- Uveitis
- Secondary Surgical Intervention to remove/Replace lens
- Pupillary Block Glaucoma IOP > 5mmHg over baseline and IOP > 25mmHg
- Corneal Edema
- Retinal Detachment
- Corneal Endothelial Cell Loss
- Secondary Glaucoma
- Hyphema
- Synechiae to Implant
- Hypopyon
- Under/Over correction
- Severe Intraocular Inflammation
- Significant Glare and/or Halos around lights
- Intraocular Infection
- Vitreous Loss

The benefit for the patient is the treatment of its cataract and improvement of his visual acuity.

Before implanting the Lucidis lens with any of the following conditions, pre-operative evaluation should be performed by a surgeon to consider the potential benefit/risk ratio.

The patients included in this observational study are planned for surgery with Lucidis lens implantation. There is no additional risk or benefit for them participating to this post-market follow-up study.




### 2 STUDY DESIGN

### 2.1 Project title

Evaluation of efficacy and long-term safety of Lucidis Lenses / PMCF.

### 2.2 Study design

This is a monocentric, longitudinal, prospective, cohort study for a population of 120 eyes on 60 to 120 patients (depending on mono or bi-lateral surgery conditions) with a cataract, receiving an Lucidis lens implant. After the cataract procedure, data collection will take place during appointments planned by the physician (after one day, one week, one month, six months and one year).

### 2.3 Investigator

Dr Kate Hashemi Institution Jules Gonin Eye Hospital / Fondation Asile des Aveugles Avenue de France 15, Lausanne, Switzerland

### 2.4 Sponsor

Dr Max Boysset - CEO SAV-IOL SA, Falaises 74, 2000 Neuchatel

#### 2.5 Facilities

Institution Jules Gonin Eye Hospital / Fondation Asile des Aveugles Avenue de France 15, Lausanne, Switzerland

### 2.6 Study duration

Provisional total duration of the study: 21 months (nine-months inclusion period + 1-year follow-up period).

All included patients will be followed up for a period of one-year nominal. The participating physicians will be given a period of nine months to enroll patients. The study will be completed as soon as the last patient included has undergone an evaluation of one year after inclusion in the study.

An interim statistical analysis will be performed after the last patient has undergone its 6 months follow-up. Data obtained from all included patients, up to the 6-months follow-up, will be used to write this interim report.




#### 3 SELECTION OF PATIENTS

#### 3.1 Patient selection method

Once the study has been initiated, the investigator will recruit the 60 to 120 patients (120 eyes) in an expected period of 6 months. The inclusion period will end at the inclusion of the last patient.

During this period, the investigator will invite all patients for whom the decision has been made to implant a Lucidis lens to take part in the study, so as to include all patients fulfilling the study inclusion criteria in a consecutive manner.

Prior to inclusion and before carrying out any study-related procedures, the investigator will first inform each patient of the study objectives, the conditions for their participation in the study, and the need to allow the study monitor to have direct access to their medical records. Patients will be given an information leaflet and informed consent form, which they are required to personally date and sign.

Before implanting the Lucidis lenses with any of the following conditions, preoperative evaluation is performed by the surgeon to consider the potential benefit/risk ratio. In case of contraindications, ie the patient already has pathologies or physiological conditions, which may be aggravated by the lens, or in cases where the lens may interfere with the possibility of examining or treating diseases, the lens will not be implanted and the patient will not be included in the study.

Additionally to exclusion criteria, the risk/benefit ratio is individually assessed for each patient with regards to safety and patient vision performance expectations. Diagnostic, anamnesis, eye biometry combined with way of life and patient expectations are considered prior the selection by the surgeon or proposal to the patient to implant a Lucidis IOL. Lucidis is an EDOF (Extended Depth Of Focus) intraocular lens that provides near and intermediate vision in addition to distance vision. Should a patient's medical status or visual expectations determined as not in adequacy with the device, alternative available devices - such as monofocal or multifocal intraocular lenses would be implanted instead. The choice of the intraocular lens based on the state of the art is an essential parameter evaluated in depth by the physician (through diagnosis, anamnesis, comorbidities, biometry, lenses optical performances, dysphotopsia, patient way of life and expectations, etc.).

#### 3.2 Selection Criteria

- adult patients (≥18 years)
- having agreed to take part in the study and complete post-operative follow-up requirements (by having signed the information leaflet-informed consent form):
- significant reduction in visual acuity and/or visual comfort from cataract;




 for whom the physician made the decision to implant a Lucidis based on medical considerations.

#### 3.3 Non-inclusion criteria

The following will not be included in the study:

- patient included in an interventional therapeutic trial at the time of inclusion;
- patient presenting contraindications for the implantation of an intraocular lens;
- patient presenting an ophthalmic disorder liable to interfere with the study endpoints;
- patient presenting with an astigmatism ≥1.0 D;
- patient refusing or unable to comply with the follow-up procedures in the study (patient unable to be reached by telephone, liable to be lost to follow-up, etc.);
- History of previous intraocular surgery in the study eye in the previous 6 months;
- patient is pregnant, breast-feeding or unable to make the decision to participate in a clinical investigation (e.g. mentally ill or handicapped person)

#### 4 PRACTICAL IMPLEMENTATION OF THE STUDY

This study does not affect the physician-patient relationship, or usual patient management. The physicians remain free in their prescribing and follow-up practices; no specific procedures or examinations are requested. The study remains within the normal treatment context.

## 4.1 Study initiation

Before the first patient is included in the study, the study protocol, case report forms and completion guidelines, the procedure for obtaining informed consent, together with the procedure for reporting adverse events will be explained to the investigator during the initiation visit.




#### 4.2 Treatment

The surgical procedures for implanting the lens are left to the discretion of the investigator according to his/her practices. All treatments administered in the context of implantation should also be reported in the "concomitant medication" section of the CRF.

#### 4.3 List of data collected

The physician will fill in a paper case report form (p-CRF) for each patient's eye, comprising:

#### 4.3.1 Data collected at inclusion:

- Date of inclusion;
- Verification of inclusion and exclusion criteria;
- Declaration by the physician that the patient has signed the information leaflet and informed consent form;
- Demographic data (age at inclusion, gender);
- Candidate eye for operation (uni- or bilateral in nature)

#### 4.3.2 Data collected at baseline visit (pre-operative):

- · Cataract history: age of onset, type of cataract;
- Pre-operative ophthalmological examination: standard slit-lamp examination, visual acuity in photopic and mesopic conditions (uncorrected visual acuity for near, intermediate (80cm), and far vision & best corrected visual acuity for far vision), contrast sensitivity and aberrometry.

#### 4.3.3 Data collected on the day of surgery:

- Operated eye
- Lens information
- General surgical procedure information (Constant value including formula biometry, type of anaesthesia, incision site). The choice of the formula is left to the discretion of the investigator. However, it shall be the same for all patients.
- Adverse event during surgery

#### 4.3.4 Data collected after surgery at day 1:

 Postoperative ophthalmological examination: standard slit-lamp examination, visual acuity in photopic and mesopic conditions (uncorrected visual acuity for near, intermediate (80cm), and far vision &




best corrected visual acuity for far vision), contrast sensitivity, aberrometry and defocus (defocus will be measured for the first 40 patients as a minimum) at the discretion of the investigator.

- Adverse events spontaneously reported by the patient;
- Specific interview concerning visual acuity, frequency of glare and halo, distorted vision.
- Possible postoperative complications
- · Change in medication intake

### 4.3.5 Data collected after surgery (at week 1, month 1, month 6, year 1):

- Postoperative ophthalmological examination: standard slit-lamp examination, visual acuity in photopic and mesopic conditions (uncorrected visual acuity for near, intermediate (80cm), and far vision & best corrected visual acuity for far vision), contrast sensitivity, aberrometry and defocus (defocus will be measured for the first 40 patients as a minimum).
- Adverse events spontaneously reported by the patient;
- Specific interview concerning visual acuity, frequency of glare and halo, distorted vision.
- Possible postoperative complications
- · Change in medication intake

#### 4.4 Evaluation schedule

The initial evaluation during the inclusion and baseline visit is done from 1 to 14 days before the date of surgery.

The evaluation schedule will then correspond as follows, for each eye:

- Day of surgery
- Day 1 (0 to 3 days after surgery)
- Week 1 (7 to 10 days after surgery)
- Month 1 (30 to 45 days after surgery)
- Month 6 (180 to 195 days after surgery)
- Year 1 (360 to 390 days after surgery).

If it is not possible to perform a visit, it must be documented and justified on the p-CRF. See also chapter 4.5 for lost patients follow-up.




In case of bilateral surgery, the Month 6 and Year 1 follow-up visits of each eye can be combined together into 1 visit, if within the timeframe. After the second eye's surgery, visual acuities are additionally measured as bilateral.




| Collected data | Screenin<br>g (study<br>inclusion | Baseline<br>visit<br>(D - 14-1) | Surgical<br>procedure<br>(D) | Follow-up Day 1<br>(D1-2) | Follow-up Week 1 (D7-10) Follow-up Month 1 (D30-45) Follow-up Month 6 (D180-195) <sup>2</sup> Follow-up Year 1 (D360-390) <sup>2</sup> |
|---|---|---|---|---|---|
| Informed consent | X | | | | |
| Demographics | Х | | | | |
| Inclusion / exclusion criteria | X | | | | |
| Candidate eye(s) for operation | Х | | | | |
| Slit lamp examination | | Х | | X1 | X |
| Cataract history | | Х | | | |
| Contrast sensitivity Photopic (85–100 lx) and Mesopic (3 lx) | | Х | | <b>X</b> <sup>1</sup> | Х |
| Uncorrected Visual Acuity – Far<br>Photopic (85–100 lx) and<br>Mesopic (3 lx) | | Х | | <b>X</b> ¹ | X |
| Uncorrected Visual Acuity –<br>Intermediate<br>Photopic (85–100 lx) and<br>Mesopic (3 lx) | | X | | X¹ | X |
| Uncorrected Visual Acuity – Near<br>Photopic (85–100 lx) and<br>Mesopic (3 lx) | | X | | X¹ | × |
| Best Corrected Visual Acuity - Far | | Х | | X1 | X |
| Defocus curve* Photopic (85–100 lx) and Mesopic (3 lx) | | Х | | X¹ | Х |
| Abberometry | | X | | X <sup>1</sup> | X |
| Operated eye | | | X | | |
| Lens information | | | Х | | |
| General surgical procedure information | | | Х | | |
| Adverse event during surgery | | | X | | |
| Adverse event spontaneously reported by patient | | | | Х | X |
| Specific interview: visual acuity,<br>frequency of glare and halo,<br>distorted vision | | | | х | X |
| Change in medication intake | | | | X | X |

<sup>\*</sup>only for the first 40 patients. In case of patient withdrawal, data will be collected on a new patient to obtain data on a minimum 40 patients, whenever possible.

## 4.5 Patients lost to follow-up

A patient will be considered lost to follow-up if s/he does not attend a scheduled visit and if the investigating physician is unable to obtain any news on the patient in the next two months after making every attempt to contact the patient.

X<sup>1</sup>: at the discretion of the investigator

<sup>&</sup>lt;sup>2</sup>: Additional follow up visits compared to standard procedure




During contact, the investigating physician will ask the patient about the reasons for not attending the scheduled visit (moved house, personal decision for example) and his/her decision regarding participation in the study and continued management.

## 4.6 End of study - withdrawal from the study

The patients will be considered to have completed the study after they have undergone a final evaluation 1 year after the inclusion visit.

The following may be considered to have withdrawn from the study:

- Patients who have requested to do so (verbal or written) via the investigator;
- patients lost to follow-up by the center, unable to be reached;
- Included patients presenting an exclusion criterion during the study (for example, inclusion in an interventional therapeutic trial).

In case of withdrawal of informed consent, non-compliance, disease progression, safety, etc. the study procedures might be stopped but the routine follow-up should be performed due to safety concerns. Data previously obtained will be retained and analyzed.

## 4.7 Monitoring

The sponsor, or an individual independent from the study and appointed by the sponsor, will perform monitoring visits, at study initiation, after one of the evaluation schedule and at study completion, as a minimum, to oversee progress in accordance with this protocol.

#### 5 ASSESSMENT METHODS

At each visit the patient will be seen by both an ophthalmologist and an optometrist. The qualified optometrist will carry out all examinations regarding visual acuity, contrast sensitivity and aberrometry. The investigating ophthalmologist will collect data through slit-lamp examination, and through interviewing the patient about any unusual sensations or adverse events based on the patient's impressions, observations and response to the question: "How are you feeling?" or "How have you felt since the last visit?". Adverse events will be recorded. An anomaly persisting at the end of the study will be monitored by the investigator until they resolve or at least stabilize.




### 6 ADVERSE EVENTS

#### 6.1 Definitions

#### 6.1.1 Definition and classification of adverse events:

An adverse event is a harmful occurrence in a person taking part in a biomedical study, whether or not this event is related to the study or study product. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the product, whether or not this is considered to be related to the use of the product (International Conference on Harmonisation, ICH).

A serious adverse event (SAE) is an event which:

- · results in death;
- is life-threatening to the person taking part in the study;
- requires inpatient hospitalization (≥ 24 hrs) or prolongation of existing hospitalization;
- results in persistent or significant disability/incapacity;
- or is a congenital anomaly/birth defect.

A life-threatening risk is an event which places the subject at immediate risk of death at the time of the event; this does not refer to an event which hypothetically may have caused death if it were more severe.

Any medically significant event which, according to the assessment based on the investigator's medical and scientific knowledge, while not immediately life-threatening, may result in the death of the patient, require inpatient hospitalization, endanger the patient, require medical or surgical intervention to prevent progression to one of the above-mentioned situations, should be perceived as serious.

Temporary transfer to a hospital outpatient clinic, an admission's department or day hospital (< 24 hrs) or inclusion in a home hospitalization system not leading to administrative hospital stay measures, is not perceived as hospitalization.

Any hospitalization occurring during a study should be reported to the sponsor by the investigator (as soon as it is brought to his/her attention).

Therefore, the following types of hospitalization are not subject to declaration: required surgical intervention planned prior to inclusion in the study, for investigations stipulated in the protocol, as a simple precautionary measure for monitoring after overdose in a patient not presenting any clinical, paraclinical or laboratory anomalies, or related to specific social circumstances affecting the patient. Any pregnancies during the study will be considered an SAE.




Unexpected adverse event: any event the nature or severity of which is not in the product instruction for use.

#### 6.1.2 Causal relationship of adverse event

The causal relationship of the adverse event should be based on the following classification:

- device related: potential imputability with the device
- surgery related: potential imputability with the surgical procedure
- other.

### 6.1.3 Severity of the adverse event

The severity of the adverse event should be based on the following classification:

- mild: generally transient, does not affect the patient's normal daily activities;
- moderate: interferes with the patient's daily activities and/or sleep;
- severe: prevents the patient's daily activities and/or sleep.

#### 6.2 Procedures

#### 6.2.1 Serious adverse events and pregnancy

Serious events are not expected in the context of this study, which is the treatment of cataract.

However, in case of serious adverse events and/or pregnancies occurring during the study, must be reported to the study sponsor by fax or mail within 24 hours of the event being notified. This report must be signed and dated by the investigator and faxed or mailed to:

Dr. Max Boysset

Fax: +41 32 566 54 01

Mail: Max Boysset <u>max.boysset@sav-iol.com</u>

and copy to:

Dr Kate Hashemi

Mail: kattayoon.hashemi@fa2.ch

Serious adverse events which have not resolved at the end of the study should be monitored by the investigator until they are resolved (or become consolidated) or until




there is evidence that there is no relationship between the event and the study conditions or until it is firmly believed that no additional information can be obtained.

#### 6.2.2 Other adverse events

Non-serious adverse events (including exacerbation of existing disorders) should be reported on the p-CRF regardless of their causal relationship, from the signing of the information leaflet and informed consent form until the end of the last study procedure.

Investigators should give their own opinion on the relation between the event and the lens implant, describe all the measures taken as a result of the event as well as the event outcome in the p-CRF.

The sponsor is responsible for the appropriate reporting of adverse events to the authorities and the Ethics Committee that approved the protocol.

### 7 DATA COLLECTION AND ANALYSIS

#### 7.1 Data collection

The investigator will receive a case report form (p-CRF) paper format for each patient for recording the evaluation results. Collected data on p-CRF will be used as source data. In case of bilateral surgery, one case report form will be completed for each eye which include bilateral visual acuity

Each patient will be assigned an identification number. The sponsor will review case report forms and collected data will be entered in Excel file at specific time (for example after monitoring visits) by an independent individual appointed by the sponsor. The entered data will be checked by another person. Then the completed cells on the Excel spreadsheet will be blocked and the document printed. The printed record must be dated and signed. The printed record will be added to the study input documentation. This file will be maintained by the sponsor who will ensure that it is valid and secure.

## 7.2 Statistical analysis

The analysis will be comparative and shall concern all patients having agreed to take part in the study. Statistical data will be evaluated for each eye, additionnaly in case of bilateral surgery visual acuity for both eyes will be analysed for each eye and together. The quantitative variables will be described in terms of sample size, mean, standard deviation, median, range and missing data. The qualitative variables will be described in terms of sample size, percentage and missing data. Two-sided 95% confidence intervals will be provided if the endpoint is considered relevant. Wilcoxon and Student significance tests will be used.




An interim statistical analysis will be performed from the 6 months data of all included patients. A final statistical analysis will be performed after the last 1-year follow-up visit of the last patient. Data will be compared to the state of the art data regarding similar lenses available on the market.

### 7.3 Required sample size

The total number of eyes to be included in the study is **120**. Indeed, based on the statistical calculations and standards described in ISO 11979-7:2018 regarding clinical investigations for ophthalmic implants, intraocular lenses, it is considered that 100 eyes would be sufficient to detect the appearance of any post-operative complications, at a statistically satisfactory rate of probability, and to discriminate the visual acuity results.




#### 8 ETHICAL AND LEGAL CONSIDERATIONS

### 8.1 Medical-regulatory framework of the study

The procedures described in this protocol, concerning the implementation, evaluation and documentation of the study are designed to ensure that the sponsor and investigating physician comply with the ethical principles defined in the Declaration of Helsinki and with the Good Clinical Practice according to the standard ISO 14155: 2011.

The study will be conducted in compliance with Swiss Law and Swiss regulatory authority's requirements and European regulatory requirements and legislation.

This observational study does not require additional biological samples of any type whatsoever, other than those normally prescribed by the physician. Except for 2 additional follow-up visits (month 6 and Year 1) and additional examination under mesopic conditions, it does not change the way in which the physician manages the patient.

### 8.2 Investigator's responsibilities

The investigator is responsible for ensuring that the study is conducted in accordance with Good Clinical Practice (GCP) guidelines as well as all the regulations governing the conduct of clinical trials in Switzerland.

Good Clinical Practice (GCP) guidelines aim to protect the rights, safety and welfare of persons taking part in research, together with the credibility and confidentiality of personal data and the study results. GCP are international standards of ethical and scientific quality concerning the development, conduct, recording and reporting of studies involving human participants.

Compliance with these reference standards provides assurance that the rights, safety, protection and well-being of patients in the study will be respected in accordance with the principles laid down in the Declaration of Helsinki, and that the clinical study data are reliable (genuine, precise and accurate).

#### 8.3 Ethics committee

The present protocol was drawn up based on the generic standard ISO 14155:2011 (Clinical investigation of medical devices for human subjects. Good clinical practice).

EU Regulation 2017/745, concerning medical devices was taken into account, together with the Federal Act on medicinal products and medical devices (Act on therapeutic products) and the ordinance on clinical trials on therapeutic products.




This study can only be undertaken after approval of the protocol and appendices has been obtained from the relevant Ethics Committee. During the study, the following documents must be submitted to the Ethics Committee for review:

- Any amendments to the protocol
- Any changes to the information leaflet and informed consent form or any document to be given to the patient.
- All cases of SAEs related to the lens implant
- · new investigator notification
- any new information concerning the safety of the device or which may interfere with the conduct of the study
- protocol deviations which may affect the results of the study.

During the study, amendments to the protocol which alter the risks and obligations of the patients, amendments and revisions made to the information leaflet and informed consent form, together with any substantial amendments must be promptly submitted to the Ethics Committee for review and approval prior to implementing any such changes.

At the end of the study, the sponsor shall notify the Ethics Committee of the end of the study, then send it the safety report, together with a summary of the study report.

#### 8.4 Patient information leaflet and informed consent form

Each patient must give his/her written informed consent after receiving a full explanation about the nature of the study. The consent form (the content of which has been approved by the Ethics Committee) must be dated and signed prior to the execution of any study-related procedures.

Before enrolment in the study, the investigator must explain the nature of the study and the consequences of their participation to the selected patients. Patients must be informed about the voluntary nature of their participation and their right to withdraw their consent at any time without affecting the quality of their future care in any way. They will be informed that alternative treatments are available should they refuse to take part in the study. Finally, they must be informed that the competent authorities and sponsor's representatives may have access to their personal study data, but that the confidentiality of this information will be respected according to current laws and regulations. The patient must be given sufficient time to read the informed consent form and to ask further questions.

After signature, a copy of the information leaflet and informed consent form will be given to the patient and a copy will be kept by the investigator on the investigation site.




The participation to the study will not generate additional cost to the patient or their health insurance. The sponsor will reimburse the additional visits based on proof of invoice for the following eligible costs:

- Outward and return trip from the place of residence to the investigator
  - o Car: 70cts / km
  - o Train: actual cost in second class
  - o Taxis: Actual costs up to a maximum of CHF 50 per trip
  - Medicalized car: costs not covered by health insurance reimbursed
  - Ambulance / not reasonably mobile: not reimbursed and/or withdrawal from the study

The cost refund by the sponsor will be made through the investigation center, the investigation center will provide the refund directly to the patient as the sponsor must not have access to patient's personal data.

### 8.5 Protection of personal data

In compliance with Swissmedic recommendations and "Swissethics" Ethics Committee Working Group guidelines, the collection and processing of data concerning the patients included in the study will only concern those data required for the implementation of the trial. The patients' names must not be communicated to the sponsor only the investigator will have access to the code. The sponsor will not have access to patient's personal data, only the patient number will be shown in the CRFs. Technical measures and appropriate organization are planned to protect personal data against unauthorized disclosure or access, destruction or accidental or unlawful alteration of data. Patients have the right to request access to their personal data through the investigator and the right to rectify any incorrect or incomplete data.

## 8.6 Premature discontinuation of the study

The sponsor or investigating physician may discontinue the study at any time. This discontinuation should take place, if possible, after mutual dialogue.

If the study were prematurely discontinued, all study materials (including data collection forms, whether completely, partly completed or blank) should be returned to the medical device company sponsoring the study.

## 8.7 Record keeping / archiving

The sponsor will register the study before carrying out the study in <a href="https://www.clinicaltrial.gov">www.clinicaltrial.gov</a>.

All study data must be archived for a minimum of 15 years after study termination or premature termination of the clinical study.

Records will be located and stored on the clinical investigation center of:
Institution Jules Gonin Eye Hospital / Fondation Asile des Aveugles




Avenue de France 15, Lausanne, Switzerland

### 8.8 Quality assurance - audit procedures

In compliance with Good Clinical Practice (GCP) guidelines, the investigating physician agrees to a possible audit by an individual whose involvement in the study is limited to this role only.

This individual is either:

- A Quality Assurance representative from the medical device company acting as the sponsor;
- An individual independent from the study and appointed by the medical device company acting as the sponsor;
- A representative from competent authorities.

At the request of medical device company acting as the sponsor, a Clinical Research Associate may also carry out random audits at the center. Quality control applies to all stages of the study, from developing the summary document to publication of the results and filing of the data used or generated in the context of the study.

### 9 USE OF RESULTS

All information and scientific data relating to the products and collected in the context of this study are considered confidential. The result of the study can be submitted (by the investigator or the sponsor) for publication or presentation to a health authority or scientific gathering without prior authorization from the investigator and the sponsor initiating the study.

### 10 FINANCIAL ASPECTS

### 10.1 Investigator fees

The sponsor will pay a fee to the investigator per surgery of 1740 CHF exc. VAT on a 120 lenses basis (total number of lenses provided).

### 10.2 Sponsor fees

The sponsor delivers 120 lenses to the investigator free of charge.




### 10.3 Additional costs

Additional costs of 10,000 CHF are accrued, including diverse professional services, publication costs, to the charge of the sponsor.




### 11 SCHEDULE

| Activities | Dates |
|---|---|
| Study start day | January 2021 – subject to ethical committee |
| | approval |
| End of enrolment | October 2021 |
| Submission of report | February 2022 |
| Use of findings (abstracts, posters, articles) | TBD |

### 12 SIGNATURES

| SAV-IOL SA, Falaises 74, 2000 Neuchâtel, | Dr Max Boysset |
|------------------------------------------|-------------------------|
| Switzerland, CHE-114.948.271 | Chief Executive Officer |

On the first hand, and

| Exercising in Institution Jules Gonin Eye | Dr Kate Hashemi Principal Investigator |
|---|---|
| Hospital / Fondation Asile des Aveugles, | |
| Avenue de France 15, Lausanne, Switzerland, | |
| CHE-109.382.412 | |

On the second hand